CLINICAL TRIAL: NCT02802683
Title: Hemodynamic Impact of Hyperbaric Versus Isobaric for Spinal Anesthesia During Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JHBahk_C/S
Record Dates: First submitted 2016-05-04; First posted 2016-06-16 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Hypotension
Keywords: Hypotension; cesarean section
MeSH Terms: conditions — Hypotension | interventions — Bupivacaine; Levobupivacaine; Phenylephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- "BUPI","P" (Experimental): patients who received hyperbaric bupivacaine and continous infusion of phenylephrine
  Interventions: Drug: Bupivacaine; Drug: Phenylephrine
- "BUPI","N" (Placebo Comparator): patients who received hyperbaric bupivacaine and continous infusion of normal saline
  Interventions: Drug: Bupivacaine; Drug: normal saline
- "LEVO","P" (Experimental): patients who received isobaric levobupivacaine and continous infusion of phenylephrine
  Interventions: Drug: Levobupivacaine; Drug: Phenylephrine
- "LEVO","N" (Active Comparator): patients who received isobaric levobupivacaine and continous infusion of normal saline
  Interventions: Drug: Levobupivacaine; Drug: normal saline

INTERVENTIONS:
Drug: Bupivacaine — spinal anesthesia with hyperbaric bupivacaine
  Other Names: Heavy bupivacaine
  Arms: "BUPI","N"; "BUPI","P"
Drug: Levobupivacaine — spinal anesthesia with isobaric levobupivacaine
  Other Names: chirocaine
  Arms: "LEVO","N"; "LEVO","P"
Drug: Phenylephrine — continous infusion of phenylephrine
  Arms: "BUPI","P"; "LEVO","P"
Drug: normal saline — continous infusion of normal saline
  Arms: "BUPI","N"; "LEVO","N"

SUMMARY:
The purpose of this study is to compare the frequency of hypotension between hyperbaric anesthetics and isobaric anesthetics during cesarean section and determine whether continuous infusion of phenylephrine is effective in mothers who received hyperbaric anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman scheduled for elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* patients who refuse involved
* patients who have pre-eclampsia
* patients who have heart disease
* patients who fetal distress is suspicious

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of hypotension events with treatment related | during 30min after spinal anesthesia
  blood pressure was obtained every 1min. A 20% decrease or more decrease in SAP compared to baseline was considered as hypotension. Hypotensive events during first 30 min was recorded as primary outcome.

SECONDARY OUTCOMES:
total dose of phenylephrine | during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bahk, Principal Investigator — Seoul National University Hospital Seoul, Korea, Republic of
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea